CLINICAL TRIAL: NCT04667663
Title: Phase Ib of Cyclophosphamide, Pomalidomide, Dexamethasone and Daratumumab (CPD-DARA) in Patients With Relapsed/Refractory Multiple Myeloma. (The CPD-DARA Study)
Brief Title: CPD-DARA in Patients With Relapsed/Refractory Multiple Myeloma.
Acronym: CPD-DARA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Janssen Pharmaceuticals (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE-19-17; 2019-004386-40 (EudraCT Number)
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Cyclophosphamide; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPD-DARA (Experimental): Drug: Daratumumab Other Name: Darzalex
  Drug: Cyclophosphamide
  Drug: Pomalidomide Other Name: Pomalyst/ Imnovid
  Drug: Dexamethasone
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab (1,800mg) will be administered by a subcutaneous injection once every week for 2 cycles (Cycles 1-2), then once every 2 weeks for 4 cycles (Cycles 3-6), and following this (Cycle 7 onwards), patients will receive daratumumab once every four weeks.
  Other Names: Darzalez
Drug: Cyclophosphamide — Cyclophosphamide will be administered PO at 50mg daily for all cohorts in the study.
Drug: Pomalidomide — Pomalidomide will be administered PO on days 1-21 of each 28 day cycle. The dose will be specified by the dose level to which the patient has been enrolled.
  Other Names: Pomalyst; Imnovid
Drug: Dexamethasone — Dexamethasone will be administered PO at 40mg on days 1, 8, 15 and 22 of each 28 day cycle.

SUMMARY:
This study is a Phase Ib, open label, single arm, adaptive multi-centre clinical study. The target population for this study are patients with relapsed/refractory multiple myeloma (MM). Patients will have a confirmed diagnosis of MM, with measurable disease as per IMWG criteria, in the second relapse and beyond (third line of therapy and beyond). Patients will need to have exposure to lenalidomide and a proteasome inhibitor. Patients will be treated with Cyclophosphamide-Pomalidomide-Dexamethasone (CPD) in combination with daratumumab (DARA) to determine the Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) of the combination.

Pomalidomide will be administered orally at three dose levels 4, 3 and 2mg on days 1-21 of each 28-day cycle. Treatment will be repeated on day 1 of a 28-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, physician's decision, or sponsor's decision to terminate the study, whichever occurs first.

DETAILED DESCRIPTION:
Primary Objective 1. To determine the MTD and RP2D for pomalidomide that can safely be administered with DARA and cyclophosphamide.

Primary Endpoint

1. To determine the incidence of DLT within the first cycle of CPD in combination with DARA at each dose level.

Secondary Objectives

1. To evaluate the safety and tolerability of the CPD-DARA regimen.
2. To evaluate efficacy measures. Secondary Endpoints

1. Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). Adverse events grade will be defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 5.0.

2. The following efficacy endpoints will be measured: i. Complete Response (CR) rate after six cycles of CPD-DARA and at the end of study treatment.

ii. Best Overall Response. iii. Minimal Residual Disease (MRD) negative rate after six cycles of CPD-DARA. iv. Progression Free Survival (PFS) and Overall Survival (OS) at 6 months and 2 years.

v. Time to Response. Exploratory Objectives

1. To assess effect of CPD-DARA treatment on patient-reported outcomes and quality of life.
2. Efficacy according to the IMWG (International Myeloma Working Group) in High Risk vs Standard Risk patients.
3. Disease Control Rate (DCR). Exploratory Endpoints

1. To assess effect of CPD-DARA treatment on patient-reported outcomes and quality of life, as assessed by the FACT-G and MyPOS questionnaires completed at study commencement, at every cycle of study treatment and at completion of the study treatment.

2. Efficacy according to the IMWG in High Risk (defined by ISS stage 3 and/or high-risk cytogenetic findings including t(4;14), t(14;16), and del17p) vs Standard Risk patients.

3. Disease Control Rate (DCR) defined as stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an informed consent form (ICF) demonstrating that he or she understands the study and all procedures involved, and confirming he or she is willing to participate.
2. Age ≥ 18 years of age.
3. Confirmed diagnosis of multiple myeloma (MM) as per IMWG Criteria (Appendix C) and measurable disease defined by the following at the time of diagnosis:

   * Monoclonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma AND
   * Measurable disease as defined by any of the following:

     * IgG multiple myeloma (MM): serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dl or urine M-protein level ≥ 200mg/24 hours;
     * IgA, IgE, IgD or IgM multiple myeloma: serum M-protein level ≥ 0.5g/dl or urine M-protein level ≥ 200mg/24 hours;
     * Light chain multiple myeloma without measurable disease in the serum or the urine:

   serum immunoglobulin free light chain ≥ 10mg/dl and abnormal serum immunoglobulin kappa lambda free light chain ratio.
4. ECOG (Eastern Cooperative Oncology Group) Performance Status ≤ 2 (Appendix B).
5. Patients with relapsed or refractory disease IMWG Criteria (Appendix C).

   • Relapsed disease (patients who achieved stable disease or better in the last line of therapy), is defined as:

   Increase of > 25% from lowest response value in any one or more of the following:
   * Serum M-component and/or (the absolute increase must be > 5 g/L)
   * Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
   * Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL
   * Bone marrow plasma cell percentage; the absolute percentage must be > 10%
   * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytoma
   * Development of hypercalcaemia (corrected serum calcium > 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder

     • Relapsed disease (in patients who have achieved CR on last line of treatment): is defined as any one of the below:
   * Reappearance of serum or urine M-protein by immunofixation or electrophoresis
   * Development of > 5% plasma cells in the bone marrow
   * Appearance of any other sign of progression (i.e., new plasmacytoma, lytic bone lesion, or hypercalcaemia) • Refractory disease (patients who failed to achieve a response [stable disease (SD) or better] to their last line of therapy).
6. Patients have received two or more prior lines of therapy (including a proteasome inhibitor and an immunomodulatory drug (IMiD)) but not more than five (induction, consolidation, ASCT maintenance is considered single line therapy for the purpose of this study). Patients with prior exposure to DARA and/or pomalidomide can also be included.
7. Patients must have pre-study laboratory results meeting the following criteria during the screening period:

   1. Haemoglobin ≥ 8 g/dL (transfusions of packed red cells are permitted to achieve this).
   2. Neutrophil count ≥ 1.5 × 10^9/L (G-CSF is permitted up to 7 days prior to screening).
   3. AST (Aspartate Transaminase) and ALT(Alanine Transaminase) ≤ 2.5 × upper limit of normal.
   4. Calculated creatinine clearance ≥ 30mL/min/1.73m2 (Cockcroft-Gault Equation; Appendix F).
   5. Platelet count ≥ 75 x 10^9/L in patients for whom <50% of bone marrow nucleated cells were plasma cells (> 50 × 109/L, otherwise).
8. Patients who are women of child-bearing potential or male partners of women of child-bearing potential must agree to use two adequate/reliable contraception methods simultaneously from signing of the informed consent form (ICF) until at least 6 months after the last study drug administration. A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months). Suitable contraceptive methods include:

   1. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable),
   3. intrauterine device (IUD) or intrauterine hormone - releasing system (IUS),
   4. bilateral tubal occlusion
   5. sexual abstinence
   6. successfully vasectomised partner
   7. the use of condoms by patients or their partners (is required even if the male patient or partner has undergone a successful vasectomy, unless the woman has had a hysterectomy).
9. Must be physically and psychologically able to undergo the treatment and adhere to the schedules outlined within this protocol.

Exclusion Criteria:

1. Life expectancy < 3 months.
2. Allogeneic stem cell transplantation at any time.
3. Autologous stem cell transplantation within 12 weeks prior to Cycle 1 Day 1.
4. Peripheral neuropathy (grade ≥ 2) as defined by the NCI CTCAE Version 5.0.
5. Meningeal or Central Nervous System (CNS) involvement of myeloma.
6. Acute or chronic active viral infections (Hep B, Hep C, HIV), systemic fungal infections and parasitic infections.
7. Acute active infection requiring antibiotics.
8. Current medical or psychiatric condition or disease that could interfere with the study procedures or results.
9. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Patients with chronic obstructive pulmonary disease (COPD) will require FEV1 testing prior to inclusion in the study.
10. Moderate or severe persistent asthma, or current uncontrolled asthma (Appendix G).
11. Diagnosis of severe chronic liver disease i.e. > stage 1 cirrhosis classified with Child-Pugh score.
12. Significant heart disease including:

    1. Myocardial Infarction within 1 year prior to registration, or unstable / uncontrolled Ischemic Heart Disease (IHD).
    2. Heart failure with NYHA (New York Heart Association) grade ≥ 2 (Appendix H).
    3. Cardiac Arrythmia (CTCAE version 5 Grade ≥ 3 or clinically significant ECG abnormalities).
    4. Screening 12 lead ECG (Electrocardiogram) showing a baseline QTcF > 470 msec.
13. Known allergy, hypersensitivity or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins or their excipients, or any of the components of the treatment regime (refer to IB/SmPC (Summary of Product Characteristics)).
14. Patients who have had any prior or concurrent invasive malignancy (other than multiple myeloma) within five years of the screening period, except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, localized prostate adenocarcinoma diagnosed ≥ 3 years and without evidence of biochemical failure, or other cancer for which the patients has undergone potentially curative therapy and has had no evidence of that disease for ≥ 10 years.
15. Patients have received an investigational drug or used an invasive medical device within 4 weeks prior to registration.
16. Patients have undergone recent major surgery within 4 weeks prior to Cycle 1 Day 1.
17. Therapeutic radiation within 14 days prior to Cycle 1 Day 1.
18. Significant malabsorption states: Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
19. Active Gastric and /or duodenal ulcer.
20. Known Amyloid Light Chain amyloidosis.
21. Contraindications to thromboprophylaxis with low molecular weight heparin (LMWH) or aspirin e.g. hypersensitivity to LMWH, history of immune-mediated heparin-induced thrombocytopenia (HIT) within the past 100 days or in the presence of circulating antibodies, active clinically significant bleeding and conditions with a high risk of haemorrhage including recent (<12 weeks (from registration) haemorrhagic stroke, gastrointestinal ulcer, presence of malignant neoplasm at high risk of bleeding, recent (< 4 weeks from registration) brain, spinal or ophthalmic surgery, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral abnormalities).
22. Vaccination with live vaccines.
23. Bone-marrow aplasia.
24. Urinary tract infection.
25. Acute urothelial toxicity from cytotoxic chemotherapy or radiation therapy.
26. Urinary outflow obstruction.
27. Patient is a woman who is pregnant, or breast-feeding, or planning to become pregnant while participating in this study or within 6 months after the last dose of any component of the treatment regimen. Or, patient is a man who plans to father a child while included in this study or within 6 months after the last dose of any component of the treatment regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT within the first cycle of CPD in combination with DARA at each dose level. | Up to cycle 1

SECONDARY OUTCOMES:
MTD for pomalidomide that can safely be administered with DARA and cyclophosphamide. | Through study treatment, an average of 1 months

OTHER OUTCOMES:
RP2D for pomalidomide that can safely be administered with DARA and cyclophosphamide. | Through study treatment, an average of 1 months

CONTACTS AND LOCATIONS:
Locations (3):
- Ireland (3):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway